CLINICAL TRIAL: NCT02549365
Title: Efficacy & Safety of Nasal Influenza Immunisation in Children - The SNIFFLE-3 Study
Brief Title: Efficacy & Safety of Nasal Influenza Immunisation in Children
Acronym: SNIFFLE-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15SM2801; 2015-003019-39 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-15 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Influenza Vaccines Efficacy and Safety
MeSH Terms: interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Administration of Live attenuated influenza vaccine (LAIV) as per national guidance. Surveillance thereafter through nasal swabbing in the event of influenza-like illness.
  Interventions: Drug: Live attenuated influenza vaccine; Procedure: Surveillance (nasal swabbing) during influenza season
- Controls (Other): Surveillance in siblings of participants in the Intervention arm, through nasal swabbing in the event of influenza-like illness, irrespective of their vaccination status.
  Interventions: Procedure: Surveillance (nasal swabbing) during influenza season

INTERVENTIONS:
Drug: Live attenuated influenza vaccine — Administration of LAIV, with subsequent surveillance (nasal swabbing) during influenza season
  Other Names: Fluenz; Flumist
  Arms: Intervention
Procedure: Surveillance (nasal swabbing) during influenza season

SUMMARY:
The UK Departments of Health now recommend annual influenza vaccination for all children 2-7 years of age, with children over 7 years eligible for vaccination if in certain higher risk clinical categories. Though data are available documenting the safety and immunogenicity of LAIV in this age group, there are little data to assess efficacy and immune correlates in UK children, and in particular atopic children. This study will enrol 200 children (and at least 200 unvaccinated household sibling controls), many with a history of asthma or recurrent wheezing, and allow an assessment of efficacy, safety and immune correlates in these children, and how this varies with prior administration of pandemic influenza vaccine and/or LAIV.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 - 18 years old
* Written informed consent from parent/guardian (or patient themselves from age 16 years), with assent from children aged 8 years and above wherever possible.

Exclusion Criteria:

* Hypersensitivity to the active ingredients, gelatin or gentamicin (a possible trace residue) [notwithstanding allergy to egg protein]
* Previous systemic allergic reaction to LAIV
* Previous allergic reaction to an influenza vaccine (not LAIV) is a relative contra-indication, which must be discussed with the site PI to confirm patient suitability
* Children/adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids**.

  **High-dose steroids is defined as a treatment course for at least one month, equivalent to a dose of prednisolone at 20mg or more per day (any age); or for children under 20kg, a dose of 1mg/kg/day or more.
* Children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.
* pregnancy
* Febrile ≥ 38.0 'C in last 72 hours
* Acute wheeze in last 72 hours requiring treatment beyond that normally prescribed for regular use by the child's treating healthcare professional
* Recent admission to hospital in last 2 weeks for acute asthma
* Current oral steroid for asthma exacerbation or course completed within last 2 weeks
* Received any blood or blood products within the past 12 weeks
* Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 276 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London / Imperial College Healthcare NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Administration of Live attenuated influenza vaccine (LAIV) as per national guidance. Surveillance thereafter through nasal swabbing in the event of influenza-like illness.
  Live attenuated influenza vaccine: Administration of LAIV, with subsequent surveillance (nasal swabbing) during influenza season
  Surveillance (nasal swabbing) during influenza season
- Controls: Surveillance in siblings of participants in the Intervention arm, through nasal swabbing in the event of influenza-like illness, irrespective of their vaccination status.
  Surveillance (nasal swabbing) during influenza season
Period: Overall Study
Arm/Group | Intervention | Controls
Started | 164 | 112
Completed | 164 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Controls | Total
Number analyzed (Participants) | 164 | 112 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 164 | 112 | 276
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 48 | 113
  Male | 99 | 64 | 163
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 164 | 112 | 276

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Efficacy
Description: Vaccine efficacy will be assessed through documentation of the incidence of laboratory confirmed influenza and other respiratory viruses in the children receiving LAIV compared to unvaccinated sibling controls
Time Frame: During 2015/2016 influenza season - precise dates to be set by Public Health England as this varies annually. Approximate duration of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Controls
Number analyzed (Participants) | 164 | 112
Participants
  Swab positive for H1N1 | 4 | 2
  Swab positive for 'flu B | 4 | 0
  Swab negative | 21 | 15
  No swab taken as not indicated | 135 | 95
Statistical Analysis 1: Comparison: Intervention vs Controls; Test type: Other; Odds Ratio (OR) = 2.89, 95% CI 2-sided [0.6 to 13.9] — Incidence of laboratory confirmed influenza is compared between those vaccinated and household controls. VE will be calculated as 1 - RR with 95% confidence intervals using Poisson regression

2. Secondary Outcome: Immune Response to LAIV
Description: To assess the immune response to vaccine and non-vaccine influenza strains before and after a single dose of LAIV administration, with respect to i. serological measures (haemagglutination inhibition titre to specific influenza strain) ii. change in specific nasal IgA responses
Time Frame: Up to 6 weeks following administration of a single dose of LAIV
Population: 39 patients provided paired blood samples pre and post LAIV 89 patients provided paired oral fluid samples pre/post LAIV
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Administration of Live attenuated influenza vaccine (LAIV) as per national guidance. Blood sample and/or oral fluid sample taken prior to, and 6 weeks post LAIV as per protocol.
Arm/Group | Intervention
Number analyzed (Participants) | 89
Participants
  >4-fold increase in HI titre to a_cal strain: number analyzed (Participants) | 39
  >4-fold increase in HI titre to a_cal strain | 1
  >4-fold increase in HI titre to a_swiss strain: number analyzed (Participants) | 39
  >4-fold increase in HI titre to a_swiss strain | 19
  >4-fold increase in HI titre to a_eng strain: number analyzed (Participants) | 39
  >4-fold increase in HI titre to a_eng strain | 4
  >4-fold increase in HI titre to b_phu strain: number analyzed (Participants) | 39
  >4-fold increase in HI titre to b_phu strain | 9
  >4-fold increase in HI titre to b_bris strain: number analyzed (Participants) | 39
  >4-fold increase in HI titre to b_bris strain | 11
  >4-fold increase in oral fluid IgA to h1 | 6
  >4-fold increase in oral fluid IgA to h3 | 19

3. Secondary Outcome: Incidence of Adverse Events (AE) and Serious Adverse Events (SAEs) in Those Received LAIV
Description: Incidence of adverse events (AE) and serious adverse events (SAEs) in children receiving LAIV, with the following sub-analyses:
  * AEs occurring up to 72 hours after LAIV in participants with a history of atopy / asthma / recurrent wheezing, compared to non-atopic participants.
  * Wheezing / asthma symptoms in subjects given LAIV who have a past medical history of asthma or recurrent wheeze in the 4 weeks prior to vaccine administration vs the 3-4 week period after LAIV.
  NB: AE data was NOT collected in household controls, as per protocol NB: AE delay not collected in Controls (as per protocol)
Time Frame: Up to 1 month after LAIV administration
Population: AE data was not collected in household controls, as per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 164
Participants
  SAE | 0
  AE | 63
  No AEFI reported | 101

ADVERSE EVENTS:
Groups:
- Intervention: Administration of Live attenuated influenza vaccine (LAIV) as per national guidance. Surveillance thereafter through nasal swabbing in the event of influenza-like illness.
  Live attenuated influenza vaccine: Administration of LAIV, with subsequent surveillance (nasal swabbing) during influenza season
  Surveillance (nasal swabbing) during influenza season
  NB: Adverse Events were not monitored/assessed for the Household "Controls"
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/164
Other Adverse Events (participants affected / at risk) | 43/164
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=164)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 27 (27)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes